CLINICAL TRIAL: NCT03235427
Title: The CAROLE (CArdiac Related Oncologic Late Effects) Study
Acronym: CAROLE
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Lucille Lee, Principal Investigator, Northwell Health
Other Study IDs: IIS-0046
Record Dates: First submitted 2017-06-06; First posted 2017-08-01 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease; Cardiac Disease; Cardiac Toxicity; Radiation; Radiation Therapy; Atherosclerotic Heart Disease; Cardiotoxicity; Breast Cancer; Lung Cancer; Lymphoma; Cancer; Carcinoma, Intraductal, Noninfiltrating
Keywords: Coronary; Coronary Disease; Coronary Arteriosclerosis; Heart Disease; Cardiotoxicity; Breast Cancer; Carcinoma; Coronary Vessels; Radiation; Radiation Therapy; Coronary Artery Disease; CAD; RT; CT; Cardiac toxicity; Cardiac calcium score; Chest RT; Lung Cancer; Lymphoma; Cardiac CT Scan; Coronary Artery; Coronary arteries; Cardiac Side Effect; Cardiac tissue; Cardiac
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Cardiotoxicity; Breast Neoplasms; Lung Neoplasms; Lymphoma; Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Coronary Disease; Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Received Radiation Therapy(RT): Patients who had received radiotherapy will be sub-stratified into those who received treatment to the left or right breast.
- Did not receive Radiation Therapy (RT): Patients who did not receive radiation treatment, but received chemotherapy, hormonal therapy, and/or surgery will be used as study controls to compare the prevalence and burden of cardiac disease as compared to radiation patients.

SUMMARY:
CAROLE seeks to evaluate the relationship between chest Radiation Therapy and coronary artery disease.

The purpose of CAROLE is to check the heart health of women who received breast cancer treatments in the past and protect them from future heart disease.

DETAILED DESCRIPTION:
Background: Within the United States, there are an estimated 3.1 million women alive who have been diagnosed with invasive breast cancer, and approximately 56% of them have received radiation. Worldwide, there are 1.4 million diagnosed annually and, in 2012, it was the most commonly diagnosed cancer in women. As patients continue to live longer, cardiac dose-related toxicity has become an issue which impacts millions globally. Guidelines are sorely needed for this large at-risk population of women.

Purpose: Radiation therapy to the chest has known cardiac late effects including coronary artery disease, fibrosis, and valvular dysfunction. Unfortunately, there is no clear evidence on which radiation doses to cardiac structures cause these late toxicities. As a result, these effects are often under-recognized until after patients have become symptomatic. More than half of breast cancer patients are treated with radiation, and many receive incidental cardiac irradiation. Many of these women also receive systemic therapy which may pose additional cardiac risks. The investigators data will help to establish baseline rates of pre-clinical and clinical disease, which can be used to inform preventative guidelines that are critically needed in this at-risk population. Additionally, the investigators data will provide a better definition of the radiation dose-relationship associated with cardiac toxicity so that it will be possible to predict more accurately who is at elevated risk for iatrogenic cardiac disease.

Research Plan: This study will identify and evaluate 200 breast cancer patients treated at the investigators institution (>6 years prior) who are at risk for treatment-related cardiac toxicity. All patients enrolled in the study will receive echocardiograms (echo), electrocardiograms (EKGs), and coronary calcium (CAC) CT scans in order to comprehensively evaluate for pre-clinical and clinical cardiac disease. Patients identified as having cardiac disease during testing will be offered referral to a cardiologist. Patients who received non-radiation treatments (chemotherapy, hormonal therapy, and/or surgery) will be compared to radiated patients to establish baseline rates of preclinical and clinical disease. Patients who received cardiotoxic systemic therapy (doxorubicin, trastuzumab, etc.) will also be evaluated in subgroup analysis. Among radiation patients, this study proposes a novel method of risk assessment, which is, to utilize a patient's stored treatment plan (from 2004-2011) and fuse it with patients current cardiac imaging to delineate an accurate dose relationship associated with clinical and pre-clinical disease. This is further described in the specific aims below:

Specific Aim 1: Identify baseline levels of clinical and pre-clinical disease in breast cancer patients.

Aim 1.1: Delineate the group of patients diagnosed and treated for breast cancer between 2004-2011, enroll health system patients with recent follow up (within 3 years).

Aim 1.2: Perform non-invasive cardiac testing (EKG, echo, CAC CT scans). Aim 1.3: Establish rates of pre-clinical and clinical disease based on pre-determined criteria.

Specific Aim 2: Create an accurate dosimetric assessment of dose to cardiac structures.

Aim 1.1: Among study patients who received radiation treatment for breast cancer, obtain stored planning CT simulation scans.

Aim 1.2: Upload CT simulation scans with dosimetric information and delineate cardiac structures at risk in order to ensure accurate and reproducible target delineation.

Aim 1.3: Fuse the CAC CT scan with the CT simulation scan to accurately assess for dose correlation between coronary calcium with the dose received.

Aim 1.4: Create a dose-relationship model for the heart and cardiac structures.

Specific Aim 3: Incorporate dosimetric cardiac risk information into the investigators institution's clinical practice, publish data, and establish updated cardiac guidelines for women who have received radiation for breast cancer.

The long-term goal of the project is to elucidate specific treatment and radiation dose-related risks, which will then be used to inform follow-up recommendations and guidelines. This project will impact the way investigators describe expected cardiac risk to patients, the way the investigators recommend follow up care, and potentially, the way the investigators prescribe treatment. At present, all patients receiving radiation for breast cancer are informed that there is a risk of cardiac late effects, however, no specific cardiac imaging or intervention is recommended other than routine medical follow up. There is little distinction given to the side of the cancer, a patient's individual anatomy, or the projected dose to the anterior heart and cardiac structures. This project will allow physicians to provide a more accurate risk profile regarding future risk of cardiac morbidity. If the study reveals a very high rate of pre-clinical atherosclerotic disease, it also may prompt more routine CAC CT screening.

ELIGIBILITY:
Inclusion Criteria:

* If you are a breast cancer survivor who was diagnosed between the ages of ≥ 18-65 years (now at age 26-78).
* It has been at least 6 years since you were diagnosed.
* If you did not have a diagnosis of heart disease before* having breast cancer.

  * (*women diagnosed with heart disease after breast cancer may still be eligible)

Exclusion Criteria:

* Patients who are unable to care for themselves or who are unable to come in for testing due to health conditions or incarceration will be rescheduled or removed in the case of chronic ineligibility. No vulnerable patient populations will be used in this study. Patients will be excluded if they have any pre-existing cardiac disease at the time of diagnosis of their breast cancer (2004-2011).
* Pregnant and nursing women are ineligible.

Ages: 26 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women aged 18-65 at the time of breast cancer diagnosis, with a minimum of 6 years since diagnosis, with no history of heart disease prior to participants breast cancer diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Multimodality Cardiology Assessment- EKG | 1 Year
  Assess whether radiation to the heart is associated with increased pre-clinical and clinical cardiac disease (as determined by a composite of multimodality cardiology assessments including EKG.
  Studies will be read using a standard, evidence based, set of criterion and documented using study templates) and compared to patients who did not receive radiation to the heart.
  All cardiac tests will be reviewed and reported as a composite with one the following; No evidence of disease/unrelated, preclinical disease, or clinical disease (non-numerically) based on the Cardiologists read of the study based on standard Pre-Specified criteria.
Multimodality Cardiology Assessment- Echocardiogram with Strain | 1 Year
  Assess whether radiation to the heart is associated with increased pre-clinical and clinical cardiac disease (as determined by a composite of multimodality cardiology assessments including Echocardiogram with Strain.
  All cardiac tests will be reviewed and reported as a composite with one the following; No evidence of disease/unrelated, preclinical disease, or clinical disease (non-numerically) based on the Cardiologists read of the study based on standard Pre-Specified criteria.
Multimodality Cardiology Assessment- Coronary Artery Calcium (CAC) CT | 1 Year
  Assess whether radiation to the heart is associated with increased pre-clinical and clinical cardiac disease (as determined by a composite of multimodality cardiology assessments including Coronary Artery Calcium (CAC) CT.
  All cardiac tests will be reviewed and reported as a composite with one the following; No evidence of disease/unrelated, preclinical disease, or clinical disease (non-numerically) based on the Cardiologists read of the study based on standard Pre-Specified criteria.

SECONDARY OUTCOMES:
Agatston Score | 1 Year
  Individual cardiac structures will be accessed using Agatston score. Agatston score is calculated using a CAC CT scan to measure for the presence of coronary artery disease based on the extent of coronary artery calcification. Specifically the left main, left anterior descending, left circumflex, and right coronary arteries are all read individually and the sum of these cardiac vessels scores is read as the overall Agatston score.
  Grading of coronary artery disease (based on total calcium score) measure is without units. Score categories are as follows: No evidence of disease/unrelated, preclinical disease, or clinical disease (non-numerically). Higher Agatston score correlates with more coronary artery disease.
  The assessment of calcium (Agatston score) on CAC CT will be compared to the dose received by the specified vessel as determined using deformable registration with prior radiation imaging (simulation CT scan).

OTHER OUTCOMES:
Composite Assessment of Cardiac Disease | 1 Year
  Sub-analysis for association of specific oncologic treatment(s) with cardiac disease (as per previously described study templates) will also be performed on patients who received multimodality treatment (RT+ chemotherapy, RT + hormonal treatment, RT+ chemo and hormonal treatment, RT + individual cardio toxic chemotherapies [anthracycline, trastuzumab, etc.]) and on different surgical approaches (lumpectomy and mastectomy). Results will be reported as a single value for each arm/group.

CONTACTS AND LOCATIONS:
Overall Officials: Lucille Lee, MD, Principal Investigator — Northwell Health; Lindsay L Puckett, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersen R, Wethal T, Gunther A, Fossa A, Edvardsen T, Fossa SD, Kjekshus J. Relation of coronary artery calcium score to premature coronary artery disease in survivors >15 years of Hodgkin's lymphoma. Am J Cardiol. 2010 Jan 15;105(2):149-52. doi: 10.1016/j.amjcard.2009.09.005. Epub 2009 Nov 14. PMID 20102909
- [Background] Correa CR, Litt HI, Hwang WT, Ferrari VA, Solin LJ, Harris EE. Coronary artery findings after left-sided compared with right-sided radiation treatment for early-stage breast cancer. J Clin Oncol. 2007 Jul 20;25(21):3031-7. doi: 10.1200/JCO.2006.08.6595. PMID 17634481
- [Background] Chang M, Suh J, Kirtani V, Dobrescu A, Haas J, Zeldis S, Shayani S, Hindenburg AA. Coronary Calcium Scanning in Patients after Adjuvant Radiation for Early Breast Cancer and Ductal Carcinoma In situ. Front Oncol. 2013 Sep 25;3:253. doi: 10.3389/fonc.2013.00253. eCollection 2013. PMID 24093087
- [Background] Santoro F, Tarantino N, Pellegrino PL, Caivano M, Lopizzo A, Di Biase M, Brunetti ND. Cardiovascular sequelae of radiation therapy. Clin Res Cardiol. 2014 Dec;103(12):955-67. doi: 10.1007/s00392-014-0718-y. Epub 2014 May 7. PMID 24803132
- [Background] Tjessem KH, Bosse G, Fossa K, Reinertsen KV, Fossa SD, Johansen S, Fossa A. Coronary calcium score in 12-year breast cancer survivors after adjuvant radiotherapy with low to moderate heart exposure - Relationship to cardiac radiation dose and cardiovascular risk factors. Radiother Oncol. 2015 Mar;114(3):328-34. doi: 10.1016/j.radonc.2015.01.006. Epub 2015 Jan 16. PMID 25600105
- [Background] Ng AK. Review of the cardiac long-term effects of therapy for Hodgkin lymphoma. Br J Haematol. 2011 Jul;154(1):23-31. doi: 10.1111/j.1365-2141.2011.08713.x. Epub 2011 May 3. PMID 21539537
- [Background] Feng M, Moran JM, Koelling T, Chughtai A, Chan JL, Freedman L, Hayman JA, Jagsi R, Jolly S, Larouere J, Soriano J, Marsh R, Pierce LJ. Development and validation of a heart atlas to study cardiac exposure to radiation following treatment for breast cancer. Int J Radiat Oncol Biol Phys. 2011 Jan 1;79(1):10-8. doi: 10.1016/j.ijrobp.2009.10.058. Epub 2010 Apr 24. PMID 20421148
- [Background] Rademaker J, Schoder H, Ariaratnam NS, Strauss HW, Yahalom J, Steingart R, Oeffinger KC. Coronary artery disease after radiation therapy for Hodgkin's lymphoma: coronary CT angiography findings and calcium scores in nine asymptomatic patients. AJR Am J Roentgenol. 2008 Jul;191(1):32-7. doi: 10.2214/AJR.07.3112. PMID 18562721
- [Background] Kim KP, Einstein AJ, Berrington de Gonzalez A. Coronary artery calcification screening: estimated radiation dose and cancer risk. Arch Intern Med. 2009 Jul 13;169(13):1188-94. doi: 10.1001/archinternmed.2009.162. PMID 19597067
- [Background] DeSantis CE, Lin CC, Mariotto AB, Siegel RL, Stein KD, Kramer JL, Alteri R, Robbins AS, Jemal A. Cancer treatment and survivorship statistics, 2014. CA Cancer J Clin. 2014 Jul-Aug;64(4):252-71. doi: 10.3322/caac.21235. Epub 2014 Jun 1. PMID 24890451
- [Background] Youlden DR, Cramb SM, Dunn NA, Muller JM, Pyke CM, Baade PD. The descriptive epidemiology of female breast cancer: an international comparison of screening, incidence, survival and mortality. Cancer Epidemiol. 2012 Jun;36(3):237-48. doi: 10.1016/j.canep.2012.02.007. Epub 2012 Mar 27. PMID 22459198
- [Background] Gyenes G, Rutqvist LE, Liedberg A, Fornander T. Long-term cardiac morbidity and mortality in a randomized trial of pre- and postoperative radiation therapy versus surgery alone in primary breast cancer. Radiother Oncol. 1998 Aug;48(2):185-90. doi: 10.1016/s0167-8140(98)00062-0. PMID 9783890
- [Background] Naghavi M, Falk E, Hecht HS, Jamieson MJ, Kaul S, Berman D, Fayad Z, Budoff MJ, Rumberger J, Naqvi TZ, Shaw LJ, Faergeman O, Cohn J, Bahr R, Koenig W, Demirovic J, Arking D, Herrera VL, Badimon J, Goldstein JA, Rudy Y, Airaksinen J, Schwartz RS, Riley WA, Mendes RA, Douglas P, Shah PK; SHAPE Task Force. From vulnerable plaque to vulnerable patient--Part III: Executive summary of the Screening for Heart Attack Prevention and Education (SHAPE) Task Force report. Am J Cardiol. 2006 Jul 17;98(2A):2H-15H. doi: 10.1016/j.amjcard.2006.03.002. Epub 2006 Jun 12. PMID 16843744
- [Background] Darby SC, Ewertz M, McGale P, Bennet AM, Blom-Goldman U, Bronnum D, Correa C, Cutter D, Gagliardi G, Gigante B, Jensen MB, Nisbet A, Peto R, Rahimi K, Taylor C, Hall P. Risk of ischemic heart disease in women after radiotherapy for breast cancer. N Engl J Med. 2013 Mar 14;368(11):987-98. doi: 10.1056/NEJMoa1209825. PMID 23484825
- [Background] Carr ZA, Land CE, Kleinerman RA, Weinstock RW, Stovall M, Griem ML, Mabuchi K. Coronary heart disease after radiotherapy for peptic ulcer disease. Int J Radiat Oncol Biol Phys. 2005 Mar 1;61(3):842-50. doi: 10.1016/j.ijrobp.2004.07.708. PMID 15708264